CLINICAL TRIAL: NCT03158272
Title: A Phase 1 Study of Cabiralizumab (BMS-986227, FPA008) Administered Alone or in Combination With Nivolumab (BMS-936558) in Advanced Malignancies
Brief Title: A Study of Cabiralzumab Given by Itself or With Nivolumab in Advanced Cancer or Cancer That Has Spread
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA025-001
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — cabiralizumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Parallel assignment will only in combination therapy arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Monotherapy (Experimental): Cabiralizumab administered as a single agent intravenous formulation
  Interventions: Biological: Cabiralizumab
- Combination Therapy (Experimental): Cabiralizumab will be administered in combination with Nivolumab as an intravenous formulation
  Interventions: Biological: Cabiralizumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Cabiralizumab — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Combination Therapy

SUMMARY:
The purpose of this study is to determine whether an investigational immuno-therapy, cabiralizumab in combination with nivolumab, is safe and tolerable in the treatment of advanced malignancies.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Performance status 0-1
* Adequate organ function
* Cohort M1, 2 and C1: Measurable disease
* Cohort M1, M2 and C1: Subjects must have histologic or cytologic confirmation of an advanced (metastatic and/or unresectable) malignant solid tumor
* Cohort C2: Documented refractory or relapsed multiple myeloma
* Subjects must be refractory to or have relapsed after standard therapies, or have no known effective treatment

Exclusion Criteria:

* Cohort M1, M2, and C1: Untreated or active central nervous system (CNS) or leptomeningeal metastases
* Cohort M1, M2, and C1: Subjects with hepatocellular carcinoma (HCC)
* Cohort C2: Subjects with solitary bone or extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Japan (4):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kamogawa-shi, Chiba
  - Local Institution, Kashiwa-shi, Chiba
  - Local Institution, Chuo-ku, Tokyo

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 participants entered the treatment period, and 19 were treated.
Groups:
- M1 Cohort: 2 mg/kg cabiralizumab monotherapy
- M2 Cohort: 4 mg/kg cabiralizumab monotherapy
- C1 Cohort: Cabiralizumab in combination with nivolumab: 4 mg/kg cabiralizumab and 3 mg/kg nivolumab in participants with solid tumor
- C2 Cohort: Cabiralizumab in combination with nivolumab: 4 mg/kg cabiralizumab and 3 mg/kg nivolumab in participants with hematologic malignancies
Period: Overall Study
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Started (Started = Entered treatment period) | 3 | 4 | 6 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 6 | 6
Not completed — Disease progression | 3 | 3 | 4 | 6
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Other reasons | 0 | 0 | 1 | 0
Not completed — Adverse event unrelated to the drug | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort | Total
Number analyzed (Participants) | 3 | 4 | 6 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (5.1) | 63.8 (7.6) | 67.0 (6.2) | 64.5 (9.4) | 65.5 (7.1)
Age, Customized [Count of Participants; unit: Participants] — Age categorization
  Participants
    <65 | 1 | 2 | 1 | 3 | 7
    >=65 | 2 | 2 | 5 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 2 | 6
  Male | 3 | 2 | 4 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 6 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 6 | 6 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) - Carbiralizumab Monotherapy
Description: The number of participants that experienced an AE during the course of the study while participating in cabiralizumab monotherapy treatment.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab monotherapy
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort
Number analyzed (Participants) | 3 | 4
Number of participants | 3 | 4

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) - Carbiralizumab Monotherapy
Description: The number of participants that experienced a SAE during the course of the study while participating in cabiralizumab monotherapy treatment.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab monotherapy
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort
Number analyzed (Participants) | 3 | 4
Number of participants | 1 | 2

3. Primary Outcome: Number of Participants With AEs Meeting Protocol-defined Dose-Limiting Toxicity (DLT) Criteria - Carbiralizumab Monotherapy
Description: The number of participants that experienced an AE meeting protocol-defined DLT criteria during the course of the study while participating in cabiralizumab monotherapy treatment.
Time Frame: 28 days (from first day of treatment)
Population: All treated participants participating in carbiralizumab monotherapy
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort
Number analyzed (Participants) | 3 | 4
Number of participants | 0 | 0

4. Primary Outcome: Number of Participants With AEs Leading to Discontinuation - Carbiralizumab Monotherapy
Description: The number of participants that experienced an AE leading to discontinuation during the course of the study while participating in cabiralizumab monotherapy treatment.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab monotherapy
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort
Number analyzed (Participants) | 3 | 4
Number of participants | 0 | 1

5. Primary Outcome: Number of Participants Who Died - Carbiralizumab Monotherapy
Description: The number of participants that died during the course of the study while participating in cabiralizumab monotherapy treatment.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab monotherapy
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort
Number analyzed (Participants) | 3 | 4
Number of participants | 0 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities - Carbiralizumab Monotherapy
Description: The number of participants that experienced a laboratory abnormality during the course of the study while participating in cabiralizumab monotherapy treatment.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab monotherapy
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort
Number analyzed (Participants) | 3 | 4
Number of participants
  HYPERCALCEMIA - grade 0 | 3 | 4
  HYPERKALEMIA - grade 0 | 2 | 4
  HYPERKALEMIA - grade 1 | 1 | 0
  HYPERNATREMIA - grade 0 | 3 | 4
  HYPOCALCEMIA - grade 0 | 3 | 2
  HYPOCALCEMIA - grade 1 | 0 | 2
  HYPOKALEMIA - grade 0 | 3 | 3
  HYPOKALEMIA -grade 1 | 0 | 1
  HYPONATREMIA - grade 0 | 1 | 4
  HYPONATREMIA - grade 1 | 2 | 0
  HEMOGLOBIN - grade 1 | 2 | 0
  HEMOGLOBIN - grade 2 | 1 | 4
  PLATELET COUNT - grade 0 | 3 | 4
  LEUKOCYTES - grade 0 | 3 | 3
  LEUKOCYTES - grade 2 | 0 | 1
  ABSOLUTE NEUTROPHIL COUNT - grade 0 | 3 | 3
  ABSOLUTE NEUTROPHIL COUNT - grade 2 | 0 | 1
  LYMPHOCYTES (ABSOLUTE) - grade 0 | 1 | 0
  LYMPHOCYTES (ABSOLUTE) - grade 2 | 2 | 3
  LYMPHOCYTES (ABSOLUTE) - grade 3 | 0 | 1
  NEUTROPHILS (ABSOLUTE) - grade 0 | 2 | 3
  NEUTROPHILS (ABSOLUTE) - grade 1 | 1 | 0
  NEUTROPHILS (ABSOLUTE) - grade 2 | 0 | 1
  CREATININE - grade 0 | 2 | 3
  CREATININE - grade 1 | 1 | 1
  ALKALINE PHOSPHATASE (ALP) - grade 0 | 0 | 3
  ALKALINE PHOSPHATASE (ALP) - grade 1 | 2 | 1
  ALKALINE PHOSPHATASE (ALP) - grade 2 | 1 | 0
  ALANINE AMINOTRANSFERASE (ALT) - grade 0 | 3 | 2
  ALANINE AMINOTRANSFERASE (ALT) - grade 1 | 0 | 2
  ASPARTATE AMINOTRANSFERASE (AST) - grade 0 | 1 | 1
  ASPARTATE AMINOTRANSFERASE (AST) - grade 1 | 2 | 1
  ASPARTATE AMINOTRANSFERASE (AST) - grade 2 | 0 | 1
  ASPARTATE AMINOTRANSFERASE (AST) - grade 3 | 0 | 1
  BILIRUBIN, TOTAL - grade 0 | 3 | 4

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) - Carbiralizumab and Nivolumab Combo Therapy
Description: The number of participants that experienced an AE during the course of the study while participating in cabiralizumab and nivolumab combination therapy.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab and nivolumab combo therapy
Measure: Number; unit: Number of participants
Arm/Group | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 6 | 6
Number of participants | 6 | 5

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) - Carbiralizumab and Nivolumab Combo Therapy
Description: The number of participants that experienced an SAE during the course of the study while participating in cabiralizumab and nivolumab combination therapy.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab and nivolumab combo therapy
Measure: Number; unit: Number of participants
Arm/Group | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 6 | 6
Number of participants | 1 | 1

9. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation - Carbiralizumab and Nivolumab Combo Therapy
Description: The number of participants that experienced an AE leading to discontinuation during the course of the study while participating in cabiralizumab and nivolumab combination therapy.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab and nivolumab combo therapy
Measure: Number; unit: Number of participants
Arm/Group | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 6 | 6
Number of participants | 1 | 1

10. Secondary Outcome: Number of Participants Who Died - Carbiralizumab and Nivolumab Combo Therapy
Description: The number of participants that died during the course of the study while participating in cabiralizumab and nivolumab combination therapy.
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab and nivolumab combo therapy
Measure: Number; unit: Number of participants
Arm/Group | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 6 | 6
Number of participants | 1 | 0

11. Secondary Outcome: Number of Participants With Laboratory Abnormalities - Carbiralizumab and Nivolumab Combination Therapy
Description: The number of participants that experienced a laboratory abnormality during the course of the study while participating in carbiralizumab and nivolumab combination therapy
Time Frame: From first dose to 30 days post last dose, assessed up to July 2019, approximately 24 months
Population: All treated participants participating in carbiralizumab and nivolumab combo therapy
Measure: Number; unit: Number of participants
Arm/Group | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 6 | 6
Number of participants
  HYPERCALCEMIA - grade 0 | 6 | 6
  HYPERKALEMIA - grade 0 | 3 | 5
  HYPERKALEMIA - grade 1 | 3 | 1
  HYPERNATREMIA - grade 0 | 6 | 5
  HYPERNATREMIA - grade 1 | 0 | 1
  HYPOCALCEMIA - grade 0 | 1 | 2
  HYPOCALCEMIA - grade 1 | 4 | 3
  HYPOCALCEMIA - grade 2 | 0 | 1
  HYPOCALCEMIA - grade 3 | 1 | 0
  HYPOKALEMIA - grade 0 | 5 | 3
  HYPOKALEMIA -grade 1 | 0 | 2
  HYPOKALEMIA - grade 3 | 0 | 1
  HYPONATREMIA - grade 0 | 3 | 5
  HYPONATREMIA - grade 1 | 3 | 1
  HEMOGLOBIN - grade 1 | 3 | 1
  HEMOGLOBIN - grade 2 | 3 | 4
  HEMOGLOBIN - grade 3 | 0 | 1
  PLATELET COUNT - grade 0 | 4 | 0
  PLATELET COUNT - grade 1 | 1 | 3
  PLATELET COUNT - grade 2 | 1 | 0
  PLATELET COUNT - grade 3 | 0 | 1
  PLATELET COUNT - grade 4 | 0 | 2
  LEUKOCYTES - grade 0 | 3 | 1
  LEUKOCYTES - grade 1 | 2 | 2
  LEUKOCYTES - grade 2 | 1 | 1
  LEUKOCYTES - grade 3 | 0 | 1
  LEUKOCYTES - grade 4 | 0 | 1
  ABSOLUTE NEUTROPHIL COUNT - grade 0 | 3 | 3
  ABSOLUTE NEUTROPHIL COUNT - grade 1 | 2 | 1
  ABSOLUTE NEUTROPHIL COUNT - grade 2 | 1 | 0
  ABSOLUTE NEUTROPHIL COUNT - grade 3 | 0 | 1
  ABSOLUTE NEUTROPHIL COUNT - grade 4 | 0 | 1
  LYMPHOCYTES (ABSOLUTE) - grade 1 | 3 | 3
  LYMPHOCYTES (ABSOLUTE) - grade 2 | 2 | 2
  LYMPHOCYTES (ABSOLUTE) - grade 3 | 1 | 1
  NEUTROPHILS (ABSOLUTE) - grade 0 | 3 | 3
  NEUTROPHILS (ABSOLUTE) - grade 1 | 2 | 1
  NEUTROPHILS (ABSOLUTE) - grade 2 | 1 | 0
  NEUTROPHILS (ABSOLUTE) - grade 3 | 0 | 1
  NEUTROPHILS (ABSOLUTE) - grade 4 | 0 | 1
  CREATININE - grade 0 | 3 | 4
  CREATININE - grade 1 | 2 | 1
  CREATININE - grade 2 | 0 | 1
  CREATININE - grade 3 | 1 | 0
  ALKALINE PHOSPHATASE (ALP) - grade 0 | 1 | 4
  ALKALINE PHOSPHATASE (ALP) - grade 1 | 3 | 2
  ALKALINE PHOSPHATASE (ALP) - grade 2 | 1 | 0
  ALKALINE PHOSPHATASE (ALP) - grade 3 | 1 | 0
  ALANINE AMINOTRANSFERASE (ALT) - grade 0 | 2 | 4
  ALANINE AMINOTRANSFERASE (ALT) - grade 1 | 4 | 1
  ALANINE AMINOTRANSFERASE (ALT) - grade 2 | 0 | 1
  ASPARTATE AMINOTRANSFERASE (AST) - grade 1 | 1 | 4
  ASPARTATE AMINOTRANSFERASE (AST) - grade 2 | 2 | 1
  ASPARTATE AMINOTRANSFERASE (AST) - grade 3 | 3 | 1
  BILIRUBIN, TOTAL - grade 0 | 5 | 6
  BILIRUBIN, TOTAL - grade 2 | 1 | 0

12. Secondary Outcome: AI_Ctrough
Description: Pharmacokinetics of cabiralizumab and nivolumab were derived from serum concentration versus time data.
  Ctrough Accumulation Index; ratio of Ctrough at steady-state (i.e. Cycle 8) to Ctrough after the first dose
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
  AI = Ctrough on cycle 8 / Ctrough on Cycle 2
Time Frame: Cycle 2 (pre-dose), Cycle 8 (pre-dose)
Population: All treated participants who completed through cycle 8 visit
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Ctrough: cycle 8 to cycle 2
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 2 | 0 | 2 | 0
Ratio of Ctrough: cycle 8 to cycle 2 | NA (NA) — Data not reported due to privacy reasons |  | NA (NA) — Data not reported due to privacy reasons |

13. Secondary Outcome: AUC(0-T)
Description: Pharmacokinetics of cabiralizumab and nivolumab were derived from serum concentration versus time data.
  AUC(0-T) is defined as the area under the serum concentration-time curve from time zero to time of last quantifiable concentration after the first dose.
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
Time Frame: Cycle 1 (from Day 1 pre-dose to Day 8, 168 hour)
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 3 | 4 | 6 | 6
h*µg/mL | 4992 (16) | 11668 (14) | 9969 (30) | 8723 (26)

14. Secondary Outcome: AUC(TAU)
Description: Pharmacokinetics of cabiralizumab and nivolumab were derived from serum concentration versus time data.
  AUC(TAU) is defined as the area under the serum concentration-time curve in one dosing interval.
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
Time Frame: Cycle 1 (from Day 1 pre-dose to Day 8, 168 hour)
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 3 | 4 | 6 | 6
h*µg/mL | 4992 (16) | 12499 (2) | 9969 (30) | 10590 (6)

15. Secondary Outcome: Cmax
Description: Pharmacokinetics of cabiralizumab and nivolumab were derived from serum concentration versus time data.
  Cmax is defined as the maximum observed serum concentration.
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
Time Frame: Cycle 1 (from Day 1 pre-dose to Day 8, 168 hour)
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 3 | 4 | 6 | 6
µg/mL | 43.7 (20) | 91.4 (7) | 84.8 (19) | 76.2 (15)

16. Secondary Outcome: Ctrough
Description: Pharmacokinetics of cabiralizumab and nivolumab were derived from serum concentration versus time data.
  Ctrough is defined as the Trough observed serum concentration (predose at each cycle).
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
Time Frame: Cycles 1, 2, 3, 4, 5, 6, 7, 8, 9
Population: All treated participants for all cohorts for Cabiralizumab;
  All treated participants for Cohorts C1 and C2 for Nivolumab.
  Note: Data reported for the cycles that were reached.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 3 | 4 | 6 | 3
µg/mL
  Cabiralizumab cycle 2 | 2.44 (105) | 18.5 (1) | 10.1 (50) | 16.5 (14)
  Cabiralizumab cycle 3: number analyzed (Participants) | 3 | 4 | 5 | 0
  Cabiralizumab cycle 3 | 4.70 (95) | 39.8 (25) | 18.8 (53) |
  Cabiralizumab cycle 4: number analyzed (Participants) | 2 | 4 | 4 | 0
  Cabiralizumab cycle 4 | 2.27 (46) | 45.8 (20) | 24.5 (48) |
  Cabiralizumab cycle 5: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cabiralizumab cycle 5 | 1.43 (64) |  | 53.3 (NA) — only 1 participant reached this cycle, CV not evaluable |
  Cabiralizumab cycle 6: number analyzed (Participants) | 2 | 0 | 1 | 0
  Cabiralizumab cycle 6 | 1.49 (88) |  | 55.8 (NA) — only 1 participant reached this cycle, CV not evaluable |
  Cabiralizumab cycle 7: number analyzed (Participants) | 2 | 0 | 2 | 0
  Cabiralizumab cycle 7 | 1.52 (108) |  | 14.0 (110) |
  Cabiralizumab cycle 8: number analyzed (Participants) | 2 | 0 | 2 | 0
  Cabiralizumab cycle 8 | 1.53 (124) |  | 37.7 (29) |
  Cabiralizumab cycle 9: number analyzed (Participants) | 1 | 0 | 1 | 0
  Cabiralizumab cycle 9 | 0.304 (NA) — only 1 participant reached this cycle, CV not evaluable |  | 30.5 (NA) — only 1 participant reached this cycle, CV not evaluable |
  Nivolumab cycle 2: number analyzed (Participants) | 0 | 0 | 6 | 3
  Nivolumab cycle 2 |  |  | 16.4 (12) | 17.5 (8)
  Nivolumab cycle 3: number analyzed (Participants) | 0 | 0 | 5 | 0
  Nivolumab cycle 3 |  |  | 25.8 (14) |
  Nivolumab cycle 5: number analyzed (Participants) | 0 | 0 | 1 | 0
  Nivolumab cycle 5 |  |  | 42.1 (NA) — only 1 participant reached this cycle, CV not evaluable |
  Nivolumab cycle 9: number analyzed (Participants) | 0 | 0 | 1 | 0
  Nivolumab cycle 9 |  |  | 49.2 (NA) — only 1 participant reached this cycle, CV not evaluable |

17. Secondary Outcome: T-HALFeff_Ctrough
Description: Pharmacokinetics of cabiralizumab and nivolumab were derived from serum concentration versus time data.
  T-HALFeff_Ctrough is defined as the effective elimination half-life that explains the degree of Ctrough accumulation observed.
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
Time Frame: Cycle 2 (pre-dose), Cycle 8 (pre-dose)
Population: All treated participants who completed through cycle 8 visit
Measure: Median (Full Range); unit: hour
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 1 | 0 | 2 | 0
hour | NA [NA to NA] — Data not reported due to privacy reasons |  | NA [NA to NA] — Data not reported due to privacy reasons |

18. Secondary Outcome: Tmax
Description: Pharmacokinetics of cabiralizumab and nivolumab were derived from serum concentration versus time data.
  Tmax is defined as the time of maximum observed serum concentration.
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
Time Frame: Cycle 1 (from Day 1 pre-dose to Day 8, 168 hour)
Population: All treated participants
Measure: Median (Full Range); unit: h (Hour)
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 3 | 4 | 6 | 6
h (Hour) | 3.18 [0.533 to 4.62] | 0.546 [0.500 to 0.633] | 1.14 [0.517 to 4.00] | 1.32 [0.550 to 4.25]

19. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA)
Description: To characterize the immunogenicity of cabiralizumab and nivolumab.
  Baseline ADA-positive participant is defined as a participant who has a ADA detected sample at baseline. ADA-positive participant is a participant with at least 1 ADA-positive sample relative to baseline after initiation of the treatment.
  Data collected from participants participating in cabiralizumab monotherapy, as well as cabiralizumab and nivolumab combination therapy.
Time Frame: Day 1 pre-dose for cycles 2, 3, 5, 9, 13, 21
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 3 | 4 | 6 | 6
Number of participants
  Cabiralizumab data | 1 | 0 | 2 | 0
  Nivolumab data | NA — No data collected for nivolumab; cohort is cabiralizumab monotherapy only | NA — No data collected for nivolumab; cohort is cabiralizumab monotherapy only | 1 | 0

20. Secondary Outcome: Best Overall Response (BOR)
Description: To assess the preliminary anti-tumor activity of cabiralizumab administered alone and in combination with nivolumab per RECIST 1.1 (M1, M2, C1 cohorts: participants with advanced solid tumors) and per IMWG criteria (Cohort C2: participants with hematologic malignancies).
  IMWG: International Myeloma Working Group
  RECIST: Response Evaluation Criteria in Solid Tumors
Time Frame: From first dose to end of follow-up, assessed up to July 2019, approximately 24 months
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 3 | 4 | 6 | 6
Number of participants
  Stable disease | 2 | 0 | 3 | 0
  Progression | 1 | 3 | 3 | 6
  Not evaluable | 0 | 1 | 3 | 0

21. Secondary Outcome: Duration of Response (DOR)
Description: To assess the preliminary anti-tumor activity of cabiralizumab administered alone and in combination with nivolumab per RECIST 1.1 (M1, M2, C1 cohorts: participants with advanced solid tumors) and per IMWG criteria (Cohort C2: participants with hematologic malignancies).
  IMWG: International Myeloma Working Group
  RECIST: Response Evaluation Criteria in Solid Tumors
  Duration of response (DOR) was listed for participants with a BOR of complete response (CR) or partial response (PR).
Time Frame: From first dose to end of follow-up
Population: All treated participants Note: there is no DOR data to report as no participant had a BOR of CR or PR or better.
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose for SAEs and AEs, assessed up to July 2019, approximately 24 months. Note: Specifically for mortality data, assessment was performed up to end of study (Apr2020 data base lock).
Groups:
- M1 Cohort: 2 mg/kg cabiralizumab monotherap
Arm/Group | M1 Cohort | M2 Cohort | C1 Cohort | C2 Cohort
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/4 | 2/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 2/6 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M1 Cohort (N=3) | M2 Cohort (N=4) | C1 Cohort (N=6) | C2 Cohort (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Gastritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M1 Cohort (N=3) | M2 Cohort (N=4) | C1 Cohort (N=6) | C2 Cohort (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1
Amylase increased (Investigations) | 1 | 2 | 4 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 6 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 4 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 3 | 6 | 4
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 3 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 2 | 4 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT03158272/SAP_000.pdf
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT03158272/Prot_001.pdf